CLINICAL TRIAL: NCT04084392
Title: Evaluating the Impact of the Bridge Clinic in Patients With Opioid Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David Marcovitz, Assistant Professor of Psychiatry, MD, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 191269
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Results first posted 2024-04-01 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Opioid Use; Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Programmatic evaluation - eligible participants will be individually randomized to either direct referral to a long-term outpatient addiction provider or referral to the Bridge Clinic while long-term outpatient addiction provider is located/identified.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Participants randomized to this arm will receive care as usual.
  Interventions: Other: Usual Care
- Bridge Clinic (Active Comparator): Participants randomized to this arm will be referred to the Bridge Clinic to facilitate identification and referral to an outpatient provider for addiction treatment.
  Interventions: Other: Bridge Clinic

INTERVENTIONS:
Other: Bridge Clinic — Referral to the Bridge Clinic for temporary outpatient addiction treatment while the bridge clinic identifies an outpatient addiction treatment provider to accept the patient for long term treatment.
  Arms: Bridge Clinic
Other: Usual Care — Referral to an outpatient provider for addiction treatment.
  Arms: Usual Care

SUMMARY:
This study aims to determine whether referral to the Bridge Clinic reduces overall index hospital length of stay when compared to direct referral to a long-term outpatient addiction provider for patients with active opioid use disorder (OUD) being considered for medications-for-addiction treatment (MAT).

ELIGIBILITY:
Inclusion Criteria:

* Inpatients at VUH with active OUD being considered for MAT.
* Patient accepting a transitional prescription for buprenorphine-naloxone or IM naltrexone whose outpatient plans are not fixed

Exclusion Criteria:

* Deemed ineligible for referral to outpatient Bridge Clinic by the Addiction Consult Team (examples include but are not limited to patients with severe, active co-occurring psychiatric disorders requiring a higher level of psychiatric care or patients for whom methadone maintenance is deemed the best choice of MAT).
* Patients previously randomized in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2022-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Marcovitz, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported will be made available (including data dictionaries) after deidentification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available 3 months following publication of outcomes and will remain available for at least 5 years.
Access Criteria: Data will be made available to researchers who provide a methodologically sound proposal that has been approved by the Vanderbilt Institutional Review Board and the study executive committee.

REFERENCES:
- [Derived] Marcovitz D, Dear ML, Donald R, Edwards DA, Kast KA, Le TDV, Shah MV, Ferrell J, Gatto C, Hennessy C, Buie R, Rice TW, Sullivan W, White KD, Van Winkle G, Wolf R, Lindsell CJ; Vanderbilt Learning Healthcare System Platform Investigators. Effect of a Co-Located Bridging Recovery Initiative on Hospital Length of Stay Among Patients With Opioid Use Disorder: The BRIDGE Randomized Clinical Trial. JAMA Netw Open. 2024 Feb 5;7(2):e2356430. doi: 10.1001/jamanetworkopen.2023.56430. PMID 38411964
- [Derived] Marcovitz DE, White KD, Sullivan W, Limper HM, Dear ML, Buie R, Edwards DA, Chastain C, Kast KA, Lindsell CJ; Vanderbilt Learning Health System Investigators. Bridging Recovery Initiative Despite Gaps in Entry (BRIDGE): study protocol for a randomized controlled trial of a bridge clinic compared with usual care for patients with opioid use disorder. Trials. 2021 Oct 30;22(1):757. doi: 10.1186/s13063-021-05698-4. PMID 34717736

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | Bridge Clinic
Started | 168 | 167
Completed | 168 | 167
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Bridge Clinic | Total
Number analyzed (Participants) | 168 | 167 | 335
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 37.9 [31.8 to 44.5] | 38.7 [32.1 to 47.0] | 38 [31.9 to 45.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 72 | 141
  Male | 99 | 95 | 194
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 159 | 161 | 320
  Unknown or Not Reported | 3 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 143 | 144 | 287
  Race: Black or African American | 20 | 16 | 36
  Race: Other | 4 | 6 | 10
  Race: Missing/Unknown | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 168 | 167 | 335

OUTCOME MEASURES:

1. Primary Outcome: Hospital Length of Stay
Description: Overall index hospital length of stay measured in days
Time Frame: approximately 3 to 42 days
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Usual Care | Bridge Clinic
Number analyzed (Participants) | 168 | 167
Hours | 232.1 (267.4) | 215.0 (236.1)

2. Secondary Outcome: Combined Cost of Index Admission and Subsequent Admissions During the Study Period
Description: Total costs, and costs for each admission and care resource used measured in dollars. This includes the cost of the index hospital admission along with any subsequent admissions during the 16-week follow up period.
Time Frame: 16 weeks post-randomization
Population: Data was missing for 24 participants.
Measure: Median (Inter-Quartile Range); unit: Dollars
Arm/Group | Usual Care | Bridge Clinic
Number analyzed (Participants) | 151 | 160
Dollars | 1705.28 [360.16 to 12146.33] | 9481.93 [1478.28 to 29376.14]

3. Secondary Outcome: Number of Participants With Successful Care Linkage
Description: Dichotomous self-reported outcome of linkage to a MAT provider as defined by attending at least one visit with a MAT provider
Time Frame: 16 weeks post-randomization
Population: Data was not available for 247 participants (136 in usual care and 111 in bridge clinic).
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Bridge Clinic
Number analyzed (Participants) | 32 | 56
Participants
  Linkage To Provider = Yes | 19 | 45
  Linkage To Provider = No | 13 | 11

4. Secondary Outcome: Number of MAT Prescriptions Filled by Participant
Description: Reported buprenorphine-naloxone (or naltrexone) prescriptions filled
Time Frame: 16 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: prescriptions filled
Arm/Group | Usual Care | Bridge Clinic
Number analyzed (Participants) | 31 | 46
prescriptions filled | 1 [0 to 6] | 10 [4 to 16]

5. Secondary Outcome: Readmissions and Emergency Department (ED) Visits
Description: Composite number of ED visits and readmissions
Time Frame: 16 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: events
Arm/Group | Usual Care | Bridge Clinic
Number analyzed (Participants) | 168 | 167
events | 0 [0 to 1] | 0 [0 to 1]

6. Secondary Outcome: Hospital and ED Free Days
Description: Days alive out of the hospital and/or ED
Time Frame: 16 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Usual Care | Bridge Clinic
Number analyzed (Participants) | 168 | 167
days | 112 [111 to 112] | 112 [107 to 112]

7. Secondary Outcome: Mortality
Description: Death in hospital or documented at 16-week follow up or in the medical record.
Time Frame: 16 weeks post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Bridge Clinic
Number analyzed (Participants) | 168 | 167
Participants | 4 | 2

8. Secondary Outcome: Recurrent Opioid Use
Description: The number of participants with recurrent opioid use.
Time Frame: 16 weeks post-randomization
Population: We were unable to assess the approximate number of times opioids were used based on the patient-reported answers provided. We were only able to determine if there was or was not recurrent opioid use.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Bridge Clinic
Number analyzed (Participants) | 32 | 56
Participants | 15 | 23

9. Secondary Outcome: Overdose
Description: Any overdose self-reported at the 16-week follow up
Time Frame: 16 weeks post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Bridge Clinic
Number analyzed (Participants) | 32 | 54
Participants | 4 | 1

10. Secondary Outcome: Quality of Life - Schwartz Outcome Scale-10 (SOS10).
Description: The Quality of Life - Schwartz Outcome Scale-10 (SOS10) survey has ten questions scored on a 0 (never) to 6 (all or nearly all of the time) scale that measures the broad domain of psychological well-being and quality of life. A total score is computed as the sum across the 10 questions. Therefore, the minimum total score is 0 (never) and the maximum score is 60 (all or nearly all of the time). Higher scores indicate greater well-being and psychological health. Therefore, higher scores are better.
Time Frame: 16 weeks post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Usual Care | Bridge Clinic
Number analyzed (Participants) | 32 | 54
score on a scale | 41.5 [32.5 to 54.25] | 47 [26 to 53.75]

11. Secondary Outcome: Opioid Use Within 30 Days
Description: Opioid use within 30 days as self-reported and assessed during the 16-week follow up phone call.
Time Frame: 30 days
Population: Data was unavailable for 303 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Bridge Clinic
Number analyzed (Participants) | 13 | 19
Participants
  No Use | 2 | 2
  Single Use | 4 | 0
  Multiple Use | 7 | 17

ADVERSE EVENTS:
Time Frame: Adverse events were tracked for each participant from study enrollment throughout the 16 week follow-up period.
Arm/Group | Usual Care | Bridge Clinic
All-Cause Mortality (participants affected / at risk) | 4/168 | 2/167
Serious Adverse Events (participants affected / at risk) | 0/168 | 0/167
Other Adverse Events (participants affected / at risk) | 0/168 | 0/167

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT04084392/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT04084392/SAP_001.pdf